CLINICAL TRIAL: NCT04307134
Title: Korean Post Marketing Surveillance Study to Observe Safety and Effectiveness of BESPONSA (REGISTERED)
Brief Title: Besponsa Post Marketing Surveillance Study
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1931027; NCT04307134 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2020-02-20; First posted 2020-03-13 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy
Keywords: Refractory and relapsed B-cell ALL
MeSH Terms: conditions — Hematologic Neoplasms; Burkitt Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- R/R ALL: Patients diagnosed as relapsed or refractory B-cell precursor lymphoblastic leukemia (ALL)
  Interventions: Drug: Inotuzumab ozogamicin

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — R/R ALL who treated with Inotuzumab ozogamicin

SUMMARY:
Besponsa is approved for the treatment of R/R B-cell ALL in Korea. In accordance with the Standards for Re-examination of New Drug, it is required to conduct a PMS. Post marketing surveillance is required to determine any problems or questions associated with besponsa after marketing in Korea, with regard to the following clauses under conditions of general clinical practice. Therefore, through this study, effectiveness and safety of besponsa will be observed.

DETAILED DESCRIPTION:
Before the approval of BESPONSA® in Korea, this non-interventional study is designated as a Post-Marketing Surveillance (PMS) Study and is a commitment to Ministry of Food and Drug Safety (MFDS), as a part of Risk Management Plan (RMP) which is required by MFDS. The safety and effectiveness information of BESPONSA® will be gathered in the setting of routine practice in Korea during the initial 6 years after the approval.

ELIGIBILITY:
Inclusion criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Patients diagnosed as relapsed or refractory B-cell precursor lymphoblastic leukemia (ALL).
2. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

1. Any patients who does not agree that Pfizer and companies working with Pfizer use his/her information.
2. Patients to whom BESPONSA® is contraindicated as per the local labeling.

   -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as relapsed or refractory B-cell precursor lymphoblastic leukemia (ALL).
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1931027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with relapsed or refractory B-cell precursor Acute Lymphoblastic Leukemia (ALL) who were prescribed Inotuzumab Ozogamicin in real world setting as a routine clinical practice across South Korea were enrolled in this study.
Groups:
- Inotuzumab Ozogamicin: Participants who were treated with Inotuzumab Ozogamicin as a part of routine clinical practice were included in this observational study. No intervention was administered under this study.
Period: Overall Study
Arm/Group | Inotuzumab Ozogamicin
Started | 108
Enrolled | 108
Treated | 107
Completed | 78
Not Completed | 30
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Other | 3
Not completed — Death | 21
Not completed — Enrolled but not Treated | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included participants who have been administered Inotuzumab Ozogamicin at least once and evaluated with safety-related outcome measures at least once.
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.21 (16.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. AEs included both SAEs and all non-SAEs. An SAE was any untoward medical occurrence in a participant administered a medicinal or nutritional product at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect or was an important medical event.
Time Frame: From first dose of study intervention (Day 1) up to 28 days post last dose of study intervention (maximum up to 311 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 107
Participants
  Participants with AEs | 99
  Participants with SAEs | 34

2. Primary Outcome: Number of Participants With Adverse Drug Reactions (ADRs) and Serious ADRs (SADRs)
Description: An ADR was any untoward medical occurrence attributed to medicinal product in participant who had received that product. SADR was an ADR that resulted in any of the following: death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect; or was an important medical event.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 107
Participants
  Participants with ADRs | 53
  Participants with SADRs | 4

3. Primary Outcome: Number of Participants With Unexpected AEs and SAEs
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. An SAE was any untoward medical occurrence in a participant administered a medicinal or nutritional product at any dose that: resulted in death; is life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect or was an important medical event. An AE was considered expected if the reported event and its specificity or severity were consistent with as pre-specified in the protocol, other than these all AEs were unexpected.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 107
Participants
  Participants with unexpected AEs | 85
  Participants with unexpected SAEs | 24

4. Primary Outcome: Number of Participants With Unexpected ADRs and SADRs
Description: An ADR was any untoward medical occurrence attributed to medicinal product in participant who had received that product. SADR was an ADR that resulted in any of the following: death; was life-threatening; required inpatient hospitalization/prolongation of hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect; or was important medical event. In this outcome measure, number of participants with unexpected ADRs and SADRs are reported. An ADR was considered expected if the reported event and its specificity or severity were consistent with as pre-specified in the protocol, other than these all ADRs were unexpected.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 107
Participants
  Participants with unexpected ADRs | 15
  Participants with unexpected SADRs | 1

5. Primary Outcome: Number of AEs According to Severity
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. AEs' severity was graded using common terminology criteria for AEs (CTCAE) version 4.0; grade 1= mild AE; grade 2= moderate AE; grade 3= severe AE; grade 4= life-threatening AE and grade 5= death.
Time Frame: as for outcome 1
Population: The safety analysis set included participants who have been administered Inotuzumab Ozogamicin at least once and evaluated with safety-related outcome measures at least once. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who had any AE and "Overall Number of Units Analyzed" signifies evaluable number of AEs.
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Number analyzed (Adverse Events) | 845
Adverse Events
  Grade 1 AEs | 252
  Grade 2 AEs | 339
  Grade 3 AEs | 179
  Grade 4 AEs | 48
  Grade 5 AEs | 27

6. Primary Outcome: Number of AEs According to Action Taken
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. Number of AEs were classified as per action taken for AEs (withdrawn [temporarily or permanently or delayed]; dose reduced; dose increased; dose not changed; unknown, and not applicable) in this outcome measure. Not applicable per protocol referred to situations if participant died or if the treatment was completed prior to the reaction/event or if drug was not administered.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Number analyzed (Adverse Events) | 845
Adverse Events
  Withdrawn (temporarily or permanently or delayed) | 46
  Dose reduced | 3
  Dose increased | 0
  Dose not changed | 319
  Unknown | 0
  Not applicable | 477

7. Primary Outcome: Number of AEs According to SAEs' Category
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. Number of AEs were classified as per SAEs category (resulted in death; is life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect and is an important medical event) in this outcome measure. One SAE could have more than 1 outcome/characteristic and have been counted in more than one category.
Time Frame: as for outcome 1
Population: The safety analysis set included participants who have been administered Inotuzumab Ozogamicin at least once and evaluated with safety-related outcome measures at least once. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who had any SAE and "Overall Number of Units Analyzed" signifies evaluable number of SAEs.
Measure: Number; unit: Serious Adverse Events
Units Other Than Participants: Serious Adverse Events
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 34
Number analyzed (Serious Adverse Events) | 60
Serious Adverse Events
  SAEs that resulted in death | 27
  SAEs that were life-threatening | 9
  SAEs that required inpatient hospitalization or prolongation of hospitalization | 45
  SAEs that resulted in persistent or significant disability/incapacity | 1
  SAEs that resulted in congenital anomaly/birth defect | 0
  SAEs that were considered as an important medical event | 0

8. Primary Outcome: Number of AEs According to Their Outcomes
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. Number of AEs were classified as per their outcomes (recovered, recovered with sequelae, recovering, not recovered, and unknown) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Number analyzed (Adverse Events) | 845
Adverse Events
  Recovered | 593
  Recovered with sequelae | 0
  Recovering | 91
  Not recovered | 153
  Unknown | 8

9. Primary Outcome: Number of AEs Based on Causality of AEs to the Study Drug
Description: AE: any untoward medical occurrence in participant administered medicinal product. Number of AEs per causality of AE to study drug (certain, probable/likely, possible, unlikely, conditional/unclassified, and not-assessable/unclassifiable) were reported. Certain: couldn't be explained by other drugs, had clinically reasonable reaction on cessation of drug and pharmacological/phenomenological reaction to drug re-administration. Probable/likely: couldn't be explained by other drugs, had clinically reasonable reaction on drug cessation. Possible: could also be explained by other drugs, lacked information/unclear information on drug discontinuation. Unlikely: not likely to have causal relationship from drug administration, could also be explained by other drugs. Conditional/unclassified: needed more data to make appropriate assessment/additional of data being reviewed. Not-assessable: lacked sufficient information/conflicting information hampering accurate causality assessment.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Number analyzed (Adverse Events) | 845
Adverse Events
  Certain | 10
  Probable/likely | 13
  Possible | 135
  Unlikely | 686
  Conditional/unclassified | 1
  Not-assessable/unclassifiable | 0

10. Primary Outcome: Number of AEs Based on Other Causality of AEs
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Number of AEs were classified as per other causality of AE to the study drug (disease under the study, other disease, concomitant treatment drug or non-drug, and others) in this outcome measure.
Time Frame: as for outcome 1
Population: The safety analysis set included participants who have been administered Inotuzumab Ozogamicin at least once and evaluated with safety-related outcome measures at least once. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who had any AE and "Overall Number of Units Analyzed" signifies number of AEs evaluable for this outcome measure.
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Number analyzed (Adverse Events) | 686
Adverse Events
  Disease under the study | 442
  Other disease | 19
  Concomitant treatment drug or non-drug | 119
  Others | 106

11. Primary Outcome: Number of Participants With AEs Classified According to Their Age at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to their baseline demographic characteristics of age (less than [<] 65 years and more than or equal to [>=] 65 years) in this outcome measure.
Time Frame: as for outcome 1
Population: The safety analysis set included participants who have been administered Inotuzumab Ozogamicin at least once and evaluated with safety-related outcome measures at least once. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who had any AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who Aged <65 years at Baseline | 82
  Participants With AEs who aged >=65 years at Baseline | 17

12. Primary Outcome: Number of Participants With AEs Classified According to Their Sex at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to their baseline demographic characteristics of sex (female and male) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who were Female | 39
  Participants With AEs who were Male | 60

13. Primary Outcome: Number of Participants With AEs Classified According to Their Diagnosis at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to their baseline demographic characteristics of diagnosis (Philadelphia [+] B-cell Acute Lymphoblastic Leukemia [ALL], Philadelphia [-] B-cell ALL, and unknown) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who had Philadelphia (+) B-cell ALL Diagnosis at Baseline | 32
  Participants With AEs who had Philadelphia (-) B-cell ALL Diagnosis at Baseline | 67
  Participants With AEs who had Unknown Diagnosis at Baseline | 0

14. Primary Outcome: Number of Participants With AEs Classified According to Their Disease Status at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily had a causal relationship with the product treatment or usage. Refractory Disease: failure to achieve complete response (CR) at the end of induction. Relapsed disease: Reappearance of blasts in the blood or bone marrow (>5%) or in any extramedullary site after a CR. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, absolute neutrophil count (ANC) > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. Number of participants with AEs were classified according to their baseline demographic characteristics of disease status (refractory, first relapsed, second relapsed and third or more relapsed) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who had Refractory Disease Status at Baseline | 9
  Participants With AEs who had First Relapsed Disease Status at Baseline | 54
  Participants With AEs who had Second Relapsed Disease Status at Baseline | 28
  Participants With AEs who had Third or More Relapsed Disease Status at Baseline | 8

15. Primary Outcome: Number of Participants With AEs Classified According to Their Renal Disorder Status at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to their baseline demographic characteristics of renal disorder status (yes or no) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who had "Yes" for Renal Disorder at Baseline | 7
  Participants With AEs who had "No" for Renal Disorder at Baseline | 92

16. Primary Outcome: Number of Participants With AEs Classified According to Their Hepatic Disorder Status at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to their baseline demographic characteristics of hepatic disorder status (yes or no) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who had "Yes" for Hepatic Disorder at Baseline | 20
  Participants With AEs who had "No" for Hepatic Disorder at Baseline | 79

17. Primary Outcome: Number of Participants With AEs Classified According to Their Allergic History Status at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to their baseline demographic characteristics of allergic history (yes or no) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who had "Yes" for Allergic history at Baseline | 49
  Participants With AEs who had "No" for Allergic history at Baseline | 50
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin; Test type: Other; p = 0.9509, Regression, Logistic — Statistical data presented based on Multiple logistic regression including Allergic history as factor and was performed to assess whether allergic history status influenced occurrence of AEs. This model produced one effect estimate for association; Odds Ratio (OR) = 999.99, 95% CI 2-sided [0.01 to 999.99]

18. Primary Outcome: Number of Participants With AEs Classified According to Their Veno-occlusive Liver Disease/ Sinusoidal Obstruction Syndrome (VOD /SOS) Status at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. VOD also known as SOS is a potentially life-threatening condition in which the small veins in the liver are blocked. This obstruction impairs blood flow through the liver and can lead to liver damage and failure. Number of participants with AEs were classified according to their baseline demographic characteristics of VOD/SOS (yes or no) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who had "Yes" for VOD/SOS status at Baseline | 0
  Participants With AEs who had "No" for VOD/SOS status at Baseline | 99

19. Primary Outcome: Number of Participants With AEs Classified According to Their Previous Systemic Therapy Status at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to their baseline demographic characteristics of previous systemic therapy status (yes, no, and unknown) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who had "Yes" for Previous Systemic Therapy at Baseline | 99
  Participants With AEs who had "No" for Previous Systemic Therapy at Baseline | 0
  Participants With AEs who had "Unknown" for Previous Systemic Therapy at Baseline | 0

20. Primary Outcome: Number of Participants With AEs Classified According to Their Previous Hematopoietic Cell Transplant Status at Baseline
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to their baseline demographic characteristics of previous hematopoietic cell transplant status (yes, no, and unknown) in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants With AEs who had "Yes" for Previous Hematopoietic Cell Transplant at Baseline | 53
  Participants With AEs who had "No" for Previous Hematopoietic Cell Transplant at Baseline | 46
  Participants With AEs who had "Unknown" for Previous Hematopoietic Cell Transplant at Baseline | 0

21. Primary Outcome: Number of Participants With AEs Classified According to Usage of Concomitant Medication Throughout the Study
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. Number of participants with AEs were classified according to the use of concomitant medications (yes and no) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) up to the end of study (maximum up to 311 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 99
Participants
  Participants with AEs who took Concomitant Medication | 99
  Participants with AEs who did not take Concomitant Medication | 0

22. Primary Outcome: Number of Elderly Participants With ADRs
Description: An ADR was any untoward medical occurrence attributed to a medicinal product in a participant who had received that product. In this outcome measure, number of elderly participants (>=65 years) with ADRs at baseline were reported.
Time Frame: as for outcome 1
Population: The safety analysis set included participants who have been administered Inotuzumab Ozogamicin at least once and evaluated with safety-related outcome measures at least once. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure who were >=65 years with any AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 17
Participants | 10

23. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: BOR was defined as the best response recorded from the start of treatment until disease progression (PD) or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. Ineffectiveness was defined as BOR of refractory disease, PD, or relapsed disease. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. Refractory Disease: failure to achieve CR at the end of induction. Relapsed disease: Reappearance of blasts in the blood or bone marrow (>5%) or in any extramedullary site after a CR.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: The effectiveness analysis set included participants who have been administered Inotuzumab Ozogamicin at least once and evaluated based upon effectiveness outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 94
Participants
  Effective | 74
  Ineffective | 20

24. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their Age at Baseline
Description: BOR was defined as the best response recorded from the start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to their baseline demographic characteristic of age (<65 years and >=65 years) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: The effectiveness analysis set included participants who have been administered Inotuzumab Ozogamicin at least once and evaluated based upon effectiveness outcome measures. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure with effective BOR.
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants with Effective BOR who Aged <65 years at Baseline | 59
  Participants with Effective BOR who Aged >=65 years at Baseline | 15
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin; Statistical data for this outcome measure is combined for all age groups in accordance with local regulations; Test type: Other; p = 0.1488, Regression, Logistic — Multiple logistic regression including age as factor; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.99 to 1.07]

25. Secondary Outcome: Number of Participants With Effective BOR Classified According to Sex at Baseline
Description: BOR was defined as the best response recorded from the start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to their baseline demographic characteristic of sex (female and male) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who were Female | 32
  Participants With Effective BOR who were Male | 42

26. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their Diagnosis at Baseline
Description: BOR was defined as the best response recorded from the start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to their baseline demographic characteristic of diagnosis (Philadelphia [+] B-cell ALL, Philadelphia [-] B-cell ALL and unknown) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who had Philadelphia (+) B-cell ALL Diagnosis at Baseline | 22
  Participants With Effective BOR who had Philadelphia (-) B-cell ALL Diagnosis at Baseline | 52
  Participants With Effective BOR who had Unknown Diagnosis at Baseline | 0

27. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their Disease Status at Baseline
Description: BOR: best response recorded from start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. Refractory Disease: failure to achieve CR at the end of induction. Relapsed disease: Reappearance of blasts in the blood or bone marrow (>5%) or in any extramedullary site after a CR. The number of participants with effective BOR were classified according to their baseline demographic characteristic of disease status (refractory, first relapsed, second relapsed and third or more relapsed) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who had Refractory Disease Status at Baseline | 8
  Participants With Effective BOR who had First Relapsed Disease Status at Baseline | 40
  Participants With Effective BOR who had Second Relapsed Disease Status at Baseline | 21
  Participants With Effective BOR who had Third or More Relapsed Disease Status at Baseline | 5

28. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their Renal Disorder at Baseline
Description: BOR: best response recorded from start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to their baseline demographic characteristic of renal disorder (yes and no) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who had Renal Disorder as "Yes" at Baseline | 4
  Participants With Effective BOR who had Renal Disorder as "No" at Baseline | 70

29. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their Hepatic Disorder at Baseline
Description: BOR: best response recorded from start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to their baseline demographic characteristic of hepatic disorder (yes and no) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who had Hepatic Disorder as "Yes" at Baseline | 17
  Participants With Effective BOR who had Hepatic Disorder as "No" at Baseline | 57

30. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their Allergic History at Baseline
Description: BOR: best response recorded from start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to their baseline demographic characteristic of allergic history (yes and no) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who had Allergic History as "Yes" at Baseline | 32
  Participants With Effective BOR who had Allergic History as "No" at Baseline | 42

31. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their VOD/SOS Status at Baseline
Description: BOR: best response recorded from start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. VOD also known as SOS is a potentially life-threatening condition in which the small veins in the liver are blocked. This obstruction impairs blood flow through the liver and can lead to liver damage and failure. The number of participants with effective BOR were classified according to their baseline demographic characteristic of VOD/SOS (yes and no) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who had VOD/SOS Status as "Yes" at Baseline | 0
  Participants With Effective BOR who had VOD/SOS Status as "No" at Baseline | 74

32. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their Previous Systemic Therapy Status at Baseline
Description: BOR: best response recorded from start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to their baseline demographic characteristic of previous systemic therapy (yes, no and unknown) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who had Previous Systemic Therapy as "Yes" at Baseline | 74
  Participants With Effective BOR who had Previous Systemic Therapy as "No" at Baseline | 0
  Participants With Effective BOR who had Previous Systemic Therapy as "Unknown" at Baseline | 0

33. Secondary Outcome: Number of Participants With Effective BOR Classified According to Their Previous Hematopoietic Cell Transplant Status at Baseline
Description: BOR: best response recorded from start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC >1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to their baseline demographic characteristic of previous hematopoietic cell transplant (yes, no and unknown) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who had Previous Hematopoietic Cell Transplant as "Yes" at Baseline | 36
  Participants With Effective BOR who had Previous Hematopoietic Cell Transplant as "No" at Baseline | 38
  Participants With Effective BOR who had Previous Hematopoietic Cell Transplant "Unknown" at Baseline | 0

34. Secondary Outcome: Number of Participants With Effective BOR Classified According to Usage of Concomitant Medication Throughout the Study
Description: BOR: best response recorded from start of treatment until PD or recurrence. Effectiveness was defined as a BOR of CR or CR with incomplete hematologic recovery. PD: Increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease. CR: No circulating blasts or extramedullary disease, trilineage hematopoiesis and < 5% blasts, ANC > 1000/microliter, platelets >100000/microliter and no recurrence for 4 weeks. CR with incomplete hematologic recovery: met all criteria for CR except platelet count and/or ANC. The number of participants with effective BOR were classified according to usage of concomitant medication (yes and no) in this outcome measure.
Time Frame: From first dose of study intervention (Day 1) until disease progression or recurrence (maximum up to 311 days)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 74
Participants
  Participants With Effective BOR who Took Concomitant Medication | 74
  Participants With Effective BOR who did not Take Concomitant Medication | 0

ADVERSE EVENTS:
Time Frame: From first dose of study intervention (Day 1) up to 28 days post last dose of study intervention (maximum up to 311 days)
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. An event may be categorized as serious in one participant and non-serious in another participant or one participant may have experienced both serious and non-serious event. The safety analysis set included participants who had been administered Inotuzumab ozogamicin at least once and evaluated with safety-related outcome measures at least once.
Arm/Group | Inotuzumab Ozogamicin
All-Cause Mortality (participants affected / at risk) | 24/107
Serious Adverse Events (participants affected / at risk) | 34/107
Other Adverse Events (participants affected / at risk) | 97/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin (N=107)
Cytopenia (Blood and lymphatic system disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Necrotising colitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Acute graft versus host disease in intestine (Immune system disorders) | 2
Acute graft versus host disease (Immune system disorders) | 1
Acute graft versus host disease in liver (Immune system disorders) | 1
Chronic graft versus host disease oral (Immune system disorders) | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1
Graft versus host disease in lung (Immune system disorders) | 1
Septic shock (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 5
Pyelonephritis acute (Infections and infestations) | 3
Bacteraemia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Enterococcal bacteraemia (Infections and infestations) | 2
Bacterial infection (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
External ear cellulitis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Cerebral infarction (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiolitis obliterans syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Venoocclusive disease (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin (N=107)
Neutropenia (Blood and lymphatic system disorders) | 29
Febrile neutropenia (Blood and lymphatic system disorders) | 28
Anaemia (Blood and lymphatic system disorders) | 19
Cytopenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Lymphopenia (Blood and lymphatic system disorders) | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2
Bicytopenia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Deafness (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Dry eye (Eye disorders) | 4
Blepharitis (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Retinal exudates (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 24
Diarrhoea (Gastrointestinal disorders) | 19
Stomatitis (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal discomfort (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Haemorrhoids (Gastrointestinal disorders) | 3
Proctalgia (Gastrointestinal disorders) | 3
Oral pain (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Oral mucosa haematoma (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Pulpless tooth (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 29
Pain (General disorders) | 5
Oedema (General disorders) | 4
Chest pain (General disorders) | 3
Chills (General disorders) | 2
Influenza like illness (General disorders) | 2
Asthenia (General disorders) | 1
Face oedema (General disorders) | 1
Generalised oedema (General disorders) | 1
Localised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholestatic liver injury (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 1
Acute graft versus host disease in skin (Immune system disorders) | 3
Acute graft versus host disease (Immune system disorders) | 2
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2
Engraftment syndrome (Immune system disorders) | 1
Graft versus host disease in lung (Immune system disorders) | 1
Graft versus host disease oral (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 10
Bacteraemia (Infections and infestations) | 8
Cytomegalovirus viraemia (Infections and infestations) | 4
Clostridium difficile colitis (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 3
Staphylococcal bacteraemia (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 2
Pneumonia fungal (Infections and infestations) | 2
Pneumonia parainfluenzae viral (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Pneumonia klebsiella (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacteriuria (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Herpes dermatitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Large intestine infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media chronic (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Pathogen resistance (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Urethral injury (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 27
Liver function test increased (Investigations) | 24
Neutrophil count decreased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 5
Blast cells present (Investigations) | 5
Blast cell count increased (Investigations) | 4
Weight increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Weight decreased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Coagulation test abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 13
Decreased appetite (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 6
Electrolyte imbalance (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemic retinopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 3
Facial paralysis (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Hydrocephalus (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Scrotal swelling (Reproductive system and breast disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 4
Hypertension (Vascular disorders) | 3
Venoocclusive disease (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT04307134/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT04307134/SAP_001.pdf